CLINICAL TRIAL: NCT06865079
Title: A Randomized, Double-blind, Placebo-controlled, 53-Week Study Evaluating the Safety and Efficacy of Intra-articular Injections of TPX-100 in Subjects With Mild to Severe Tibio- Femoral Osteoarthritis of the Knee
Brief Title: 53-Week Study Evaluating the Safety and Efficacy of Intra-articular Injections of TPX-100 With Mild to Severe Tibio-Femoral Osteoarthritis of the Knee
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OrthoTrophix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPX-100-6
Record Dates: First submitted 2025-02-25; First posted 2025-03-07 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis (OA) of the Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clinical Research Organizations (CROs) Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TPX-100 (200 mg per dose) (Experimental): TPX-100 (200 mg per dose) for intra-articular injection administered once-weekly (Week 1, 2, 3 and 4) to a single target knee of the subject for 4 injections.
  Interventions: Drug: TPX-100 200mg, Once weekly for 4 weeks
- Placebo / PBS (Placebo Comparator): PBS placebo for intra-articular injection administered once-weekly (Week 1, 2, 3 and 4) to a single target knee of the subject for 4 injections.
  Interventions: Other: PBS

INTERVENTIONS:
Drug: TPX-100 200mg, Once weekly for 4 weeks — TPX-100 (200 mg per dose) will be administered once-weekly (Week 1, 2, 3 & 4) to a single target knee of the subject for 4 injections.
  TPX-100 can be administered by conventional methods such as subcutaneous or intra-articular injection.
  Arms: TPX-100 (200 mg per dose)
Other: PBS — PBS / placebo for intra-articular injection administered once-weekly (Week 1, 2, 3 and 4) to a single target knee of the subject for 4 injections
  Arms: Placebo / PBS

SUMMARY:
53-Week Study Evaluating the Safety and Efficacy of Intra-articular (IA) Injections of TPX-100 vs Placebo in Subjects with Mild to Severe Tibio-Femoral Osteoarthritis of the Knee

DETAILED DESCRIPTION:
This multicenter, double-blind, placebo controlled, randomized study is designed to investigate the safety and efficacy of TPX-100 administered in 4 weekly doses of 200 mg per dose in subjects with tibio-femoral osteoarthritis. The B-score as determined by MRI analysis is the final inclusion criteria, which will be determined by MRI-based assessment. A standardized screening MRI will be obtained on otherwise eligible candidates.

For enrolled subjects, the Screening MRI will serve as the Baseline MRI. Enrolled subjects will be assigned randomly to receive either TPX-100 or PBS placebo, 4 weekly IA injections administered into the target knee by fluoroscopy or ultrasound guidance.

Subjects will undergo follow-up knee MRIs at Week 27 and Week 53 after the first injection. All MRIs will be read by computer-based, standardized methods, blind to treatment assignment and temporal sequence, to provide the imaging outcome measures. Subjects will complete PROs at Week 1 (Baseline), Week 27 and Week 53. A clinical safety evaluation will be performed at Week 13, and a safety tele-visit or telephone call will be performed at Week 36. Adverse events, regardless of causation, and concomitant medications will be documented at all study visits and at the Week 37 tele-visit/telephone call. Clinical laboratory assessments will be obtained at Screening, Baseline (Week 1), and Weeks 2, 3, 4; and at the in-person follow up visits.

All enrolled subjects will be assigned randomly to receive either TPX-100 or PBS placebo, in 4 weekly IA injections administered into the target knee by fluoroscopy or ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria

Volunteers will be included in the study only if they satisfy all the following criteria:

1. Able to read, understand, sign, and date the subject informed consent.
2. Have given written informed consent before any study-related activities are carried out and are able to understand the nature and purpose of the trial, including possible risks and adverse effects.
3. Adult males and females, 50 to 80 years of age (inclusive) at Screening.
4. Body weight less than 136 kgs (300 lbs) at Screening.
5. Except for OA, subject is medically healthy (in the opinion of the PI), as determined by prestudy medical history, and without clinically significant abnormalities including:

   1. Clinically relevant findings on physical examination that would preclude trial compliance.
   2. Heart rate <40 BPM or >100 BPM after 5 minutes rest in supine or semi-supine position.
   3. Body temperature <95.9°F or >99.8°F. Note: The above assessments may be repeated, if abnormal values are recorded in the first instance, at the discretion of the Investigator (or delegate).
6. Available X-Ray of target knee obtained within 12 months prior to Screening with radiographic evidence of osteoarthritis in the medial and/or lateral tibio-femoral compartment; KL grading is not required.
7. Clinical diagnosis of knee OA with at least 2 of the 4 following signs/symptoms in the target knee, and in the absence of palpable warmth suggesting synovitis or infection:

   * Crepitus on knee extension
   * Bony tenderness
   * Bony enlargement
   * Morning stiffness in target knee <30 minutes
8. Stability of Cruciate and collateral ligaments as defined by clinical examination (e.g. tests such as Lachman, pivot shift, posterior drawer, posterior sag, valgus and Varus stress).
9. Results of the KOOS Knee Survey Screening Questionnaire performed at Screening for the target knee that indicate either: moderate or greater difficulty in at least 5 of 17 questions (A1-17) in the "Function, daily living" subsection; or a total score of at least 20/68 in that subsection.
10. Results of the KOOS Knee Survey Screening Questionnaire performed at Screening that indicate moderate or greater pain on question P6 "pain going up or down stairs" in the target knee.
11. Willing to use only acetaminophen (Tylenol® or equivalent), hydrocodone, orhydrocodone/acetaminophen (e.g., Norco® or equivalent) for breakthrough pain during the4-week injection period. The maximum dose of acetaminophen from all sources must not exceed 4000 mg/day.
12. Willing NOT to use non-steroidal anti-inflammatory drugs such as aspirin, ibuprofen (Motrin® or equivalent), or naproxen (Aleve® or equivalent) during the 4-week injection period.
13. Willing NOT to use approved or investigational IA products for knee OA for the duration of participation in the study.
14. If using GLP-1 medications such as Wegovy® or similar, must be on a stable dose for at least 2 months prior to Screening.
15. Female subjects of childbearing potential who are sexually active (non-abstinent) must agree to and comply with using 2 highly effective methods of birth control (oral contraceptive implant, injectable or indwelling intrauterine device, condom with spermicide or sexual abstinence) while participating in the study. Male participants must agree to use a barrier contraception method to prevent pregnancy, and agree not to donate sperm from the time of the first injection through the end of the study.
16. Willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.
17. MRI Screening: Tibio-femoral osteoarthritis with MRI based femoral B-score at Screening of 0.5 or greater in at least one knee as determined by central analysis.

Exclusion Criteria

Subjects are excluded from the study if any of the following criteria are met:

1. Contraindication to MRI.
2. Demonstrated clinically significant (required intervention, e.g., emergency room visit, epinephrine administration) allergic reactions (e.g., food, drug, or atopic reactions, asthmatic episodes) which, in the opinion of the Investigator, would interfere with the volunteer's ability to participate in the trial.
3. Prior surgery in the target knee, excluding procedures for debridement only (no previous micro-fracture procedure).
4. Knee joint replacement or any other knee surgery planned in either knee while participating in the study.
5. Moderate or severe pain in the contralateral (non-target) knee.
6. History of fibromyalgia, rheumatoid arthritis (RA), psoriatic arthritis, or any other autoimmune or infectious cause for arthritis; or referred knee pain from hip or spinal disease.
7. Knee effusion >2+ on the following clinical scale:

   1. Zero = No wave produced on down stroke
   2. Trace = Small wave on medial side with down stroke
   3. 1+ = Larger bulge on medial side with down stroke
   4. 2+ = Effusion spontaneously returned to medial side after upstroke (no down stroke necessary)
   5. 3+ = So much fluid that it was not possible to move the effusion out of the medial aspect of the knee
8. Last viscosupplementation (e.g., Synvisc® or similar hyaluronic acid product) injected into either knee < 3 months before Screening.
9. Last IA injection of corticosteroids < 2 months before Screening.
10. Current (within previous month before Screening) of use of any systemic steroids (except inhaled corticosteroids for allergy or respiratory problems).
11. Known hypersensitivity to any of the study drug ingredients.
12. Known hypersensitivity to acetaminophen or hydrocodone.
13. History of arthroscopy in the target knee in the 3 months before Screening.
14. History of septic arthritis, gout, or pseudo-gout in either knee in the year before Screening.
15. Clinical signs in the opinion of the Investigator of acute meniscal tear (e.g. locking or acute mechanical signs or symptoms consistent with meniscal tear) in either knee.
16. Skin lesion, rash, infection, or hypersensitivity in the target knee at or near the injection site at Screening.
17. Bleeding problems, platelet or coagulation deficiency that, in the option of the Investigator, contraindicates IA injection.
18. Active systemic infection at Screening or immediately pre-dose on any IA injection day, including chronic viral infection.
19. Current treatment or treatment within 2 years prior to Screening for any malignancy except basal cell or squamous cell carcinoma of the skin, prostate or cervical cancer in situ, unless with specific written permission provided by the Sponsor's Medical Monitor.
20. Women of childbearing potential who are pregnant, nursing, or planning to become pregnant, and women or men who do not agree to remain on an acceptable method of birth control throughout the entire study period.
21. Participation in other clinical OA drug studies within 1 year prior to Screening except epidemiologic studies involving no drug treatment.
22. Any participation in other clinical OA stem cell or gene therapy studies.
23. Currently taking paclitaxel (mitotic inhibitor), natalizumab (anti-integrin monoclonal antibody), or any other anti-integrin treatment.
24. Routine consumption of more than 3 alcoholic drinks a day (definition of 1 alcoholic drink:

    * 12-ounces of beer, 8-ounces of malt liquor, 5-ounces of wine, 1.5- ounces or a "shot" of 80-proof distilled spirits or liquor such as gin, rum, vodka, or whiskey).
25. History of substance abuse in the opinion of the Investigator within the two years prior to Screening.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2027-05-25 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Toxicity Reaction (CTC 5.0 standard） | Baseline to Study Week 27 and Study Week 53
  CTC 5.0, also known as Common Terminology Criteria for Adverse/Serious Adverse Events version 5.0, is an extensively used classification system for assessing drug toxicity. This system categorizes drug toxicity into five levels: Grade 0, Grade 1, Grade 2, Grade 3, and Grade 4.

SECONDARY OUTCOMES:
Change in Physical Function & Pain of the Target Knee | Baseline to Study Week 27 and Study Week 53
  The Western Ontario and MacMaster Universities Osteoarthritis Index (WOMAC®) evaluation scales will be utilized to evaluate patient progression or benefit.
  WOMAC® is widely used in the evaluation of Knee Osteoarthritis. It is a patient self-administered questionnaire consisting of 24 items divided into 3 subscales:
  * Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright
  * Stiffness (2 items): after first waking and later in the day
  * Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties
Change in MRI-based femoral B-score which ranges from -2 to +7, with higher scores indicating greater severity | Baseline to Study Week 27 and Study Week 53
  To evaluate structural changes in subchondral bone in IA TPX-100-treated versus IA placebo-exposed knees.
To evaluate Pain Frequency in the Target Knee by KOOS evaluation of question 1 which ranges from 0 (Never) - 4 (Always). | Baseline to Study Week 27 and Study Week 53
  Evaluation of the frequency of pain in the target knee will be evaluated by the KOOS pain scale in which question 1 will be evaluated. Knee injury and Osteoarthritis Outcome Score (KOOS) is an extension of the WOMAC Osteoarthritis Index with the purpose of evaluating short-term and long-term symptoms and function in subjects with knee injury and osteoarthritis. The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn McGuire - Chief Medical Officer, M.D. FAAN, Study Chair — OrthoTrophix, Inc
Locations (33):
- United States (33):
  - Elite Clinical Network, Scottsdale, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Legent Orthopedic Hospital, Carrolton, California
  - Medvin Clinical Research, Covina, California
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Marvel Clinical Research (Elite Clinical Network), Huntington Beach, California
  - Medvin Clinical Research Center, Riverside, California
  - Medvin Clinical Research Center, Tujunga, California
  - Medvin Clinical Research Center, Whittier, California
  - K2 Medical Research, Maitland, Florida
  - Wellness Research Center, Miami, Florida
  - Well Pharma Medical Research, Miami, Florida
  - Las Mercedes Medical Research, Miami, Florida
  - Drug Studies of America, Marietta, Georgia
  - AMR Kansas City, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - AMR Lexington, Lexington, Kentucky
  - Accurate Clinical Research Inc., Lake Charles, Louisiana
  - Mayo Clinic (Rochester), Rochester, Minnesota
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Hightower Clinical, Oklahoma City, Oklahoma
  - University Orthopedics Center, Altoona, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - AMR Knoxville, Knoxville, Tennessee
  - Accurate Clinical Research, LLC, Baytown, Texas
  - Texas Orthopedic Specialist, Bedford, Texas
  - First Surgical Hospital, Bellaire, Texas
  - Accurate Clinical Research, Houston, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - CenExel, Salt Lake City, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah